CLINICAL TRIAL: NCT07209488
Title: Evidence-based Modeling for Acquired Dyslexia Treatments
Brief Title: Acquired Dyslexia Modeling and Treatment
Acronym: AMT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, William W. Graves, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2025001100; R56DC022256 (NIH)
Record Dates: First submitted 2025-10-02; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Stroke; Dyslexia, Acquired
Keywords: reading; computational model; treatment; therapy
MeSH Terms: conditions — Stroke; Dyslexia, Acquired

STUDY DESIGN:
Intervention Model Description: The study model is a partial crossover design in that participants receiving model-matched therapy will continue with the same therapy in the 2nd half of the study, while those receiving the non-model-matched therapy will be switched in the 2nd half to the other therapy.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Model-matched (Experimental): This group will receive the therapy, either phonological or semantics-based, that matches the computational model prediction for the source of their reading impairment. They will receive this for the first 60 total hours of therapy, and for the second 60 hours of therapy.
  Interventions: Behavioral: Phono-Motor Therapy; Behavioral: Semantic Feature Analysis
- Model-non-matched (Active Comparator): This group will receive the therapy, either phonological or semantics-based, that does not match the computational model prediction for the source of their reading impairment. They will receive this for the first 60 total hours of therapy. For the second 60 hours, they will receive the other therapy.
  Interventions: Behavioral: Phono-Motor Therapy; Behavioral: Semantic Feature Analysis

INTERVENTIONS:
Behavioral: Phono-Motor Therapy — Orthographic stimuli (letters) are introduced from the beginning as each phoneme is being trained. This maintains the focus on phonology, while emphasizing its relevance to reading. PMT consists of an initial phase focused on training of individual phonemes and phoneme sequences in spoken language, followed by written language tasks. English phonemes are first trained in isolation, followed by phoneme sequences in words and pseudowords. They are trained multi-modally through emphasis on auditory, motor, tactile-kinesthetic, visual, and orthographic representations for each consonant and vowel. When sequences are introduced, focus on phonology is maintained by training on pseudowords first before real words are introduced. Participants work on identifying, repeating, parsing, blending, and manipulating phonemes that make up the pseudoword and word stimuli. To maintain focus on phonology, pictures and definitions of the stimuli are never shown or discussed.
  Other Names: PMT
Behavioral: Semantic Feature Analysis — SFA activates semantic features of the target word to help retrieve the spoken form of the word. To target reading, a modified SFA is used with written words rather than pictures as the primary materials. Pictures are instead included for each word as a semantic feature. Stimuli will consist of 80 highly imageable nouns with a range of word frequencies. During treatment the therapist will present a written noun and ask the participant a series of questions about the features of that noun. For example, if the presented noun is "juice", the therapist would have the participant select the corresponding picture from an array of pictures. The therapist then would ask, "what do you do with it?" (eliciting a feature from the "function" category) and "where do you store it in your home?" (eliciting a feature from the "context" category). This is done for a total of 6 categories of semantic features. The process is repeated until the participant reads the noun correctly three times in a row.
  Other Names: SFA

SUMMARY:
This study is a low-risk, early phase 1, multicenter trial to test the use of a computational (neural network) cognitive model of reading to simulate acquired dyslexia and its treatment. The aim is to determine whether there is an advantage to receiving the treatment the model predicts to be advantageous compared to the alternative treatment. All participants will receive two full rounds of treatment. A round of treatment will consist of either phonomotor treatment (PMT) or semantic feature analysis (SFA) for 60 hours, distributed over 5 days a week for 2 hours a day.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English as a first language pre-stroke by self report.
* Normal or corrected-to-normal vision.
* Normal or aided hearing.
* Left hemisphere ischemic or hemorrhagic stroke (as verified by a structural brain scan).
* Impaired reading as confirmed by significant impairment in the Basic Skills cluster of the Woodcock Reading Mastery Test - III.

Exclusion Criteria:

* Diagnosed pre-stroke neurological disease affecting the brain other than left hemisphere stroke.
* Severe apraxia of speech (determined by consensus judgment among speech-language pathologists).
* History of learning disabilities such as developmental dyslexia or current self-reported major psychiatric disorders.
* Inability to undergo, or provide a copy of, a post-stroke brain imaging scan.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants in the study population will be given equal consideration for inclusion, and no preference will be given on the basis of gender. This measure is based on self-representation of gender identity.
Enrollment: 12 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Woodcock Reading Mastery Test - III | Baseline, following the first 60 hours of therapy, and following the final 60 hours of therapy.
  The WRMT-III is a standardized measure of reading skills.
Test words and pseudowords | Baseline, following the first 60 hours of therapy, and following the final 60 hours of therapy.
  Change in accuracy of reading 120 test words and 80 pseudowords

SECONDARY OUTCOMES:
Western Aphasia Battery - Revised | Baseline, following the first 60 hours of therapy, and following the final 60 hours of therapy.
  The WAB - R is a standard measure of aphasia severity. It determines both the degree of aphasia and whether treatment has any impact on aspects of aphasia other than acquired dyslexia.
Comprehensive Aphasia Test - Disability Quotient | Baseline, following the first 60 hours of therapy, and following the final 60 hours of therapy.
  The CAT - DQ is a self-report measure of subjectively perceived degree of disability.

CONTACTS AND LOCATIONS:
Overall Officials: William W Graves, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (3):
- United States (3):
  - Florida State University, Tallahassee, Florida
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Kessler Foundation, West Orange, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Pursuant to the rules of the Institutional Review Board of Rutgers, The State University of New Jersey, only data that can be fully de-identified will be shared. All data collected using non-proprietary (non-copyrighted) instruments are expected to be de-identifiable and therefore will be shared in de-identified form. These include: structural brain images (de-faced), results of the test for hemi-spatial neglect, the experimental list of 120 words and 80 pseudowords for reading aloud, and results of touch-screen choice tasks for testing phonological, semantic, and orthographic knowledge.
Supporting Information: Study Protocol
Time Frame: We will make the behavioral and brain MRI data available through the Open Science Framework (OSF) repository as soon as possible, and no later than the time of an associated publication or end of the performance period, whichever comes first. We will also make the data available for as long as we anticipate it being useful for the larger research community, institutions, and/or the broader public.
Access Criteria: Access will be freely available by anyone using the OSF.